CLINICAL TRIAL: NCT04575051
Title: HearCARE: Hearing for Communication and Resident Engagement
Brief Title: Hearing for Communication and Resident Engagement
Acronym: HearCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Catherine Palmer, Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY19120233; HL-2019C1-16067 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2020-09-21; First posted 2020-10-05 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-10

CONDITIONS: Hearing Loss, Age-Related
Keywords: hearing loss, communication, social participation
MeSH Terms: conditions — Presbycusis; Hearing Loss; Communication

STUDY DESIGN:
Intervention Model Description: Open cohort stepped-wedge cluster randomized design with a phased, randomized roll out
Who Masked: Outcomes Assessor
Masking Description: The data collectors will be masked to which phase the facility is in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HearCARE (Consult+Engage) (Active Comparator): Residents will be exposed to the Consult Model and the Engage Model.
  Interventions: Other: Consult Model; Other: Engage Model
- Consult Model (Other): The Consult Model (i.e., usual care) is an acute care strategy, relying on a monthly Audiologist visit to the facility.
  Interventions: Other: Consult Model

INTERVENTIONS:
Other: Consult Model — The Consult Model (i.e., usual care) is an acute care strategy, relying on a monthly Audiologist visit to the facility.
Other: Engage Model — The Engage Model is a chronic care approach to supportive hearing loss self-management of ARHL. Engage includes (a) hearing screening for all residents, (b) an individualized communication plan for those with an identified hearing loss (e.g., one-to-one, group, telephone, television plans, hearing aid trouble shooting, communication strategies, etc.), (c) provision of simple, non-custom amplifiers, (d) referral to audiology if needed, and (e) ongoing support provided by trained personnel (Communication Facilitator) under the supervision of the audiologist.
  Arms: HearCARE (Consult+Engage)

SUMMARY:
Amplification is a well-established, evidence-based front-line treatment for those with impaired communication secondary to Age Related Hearing Loss (ARHL). ARHL is the most prevalent cause of communication impairment among older adults. The challenge in treating ARHL is identifying a care model that effectively promotes adherence to individualized-treatment recommendations allowing the end-user to self-manage hearing loss with appropriate support. This proposal compares the two most common models of care for ARHL provided to adults in assisted living/personal care communities. The Consult Model (i.e., usual care) is an acute care strategy, relying on a monthly Audiologist visit to the facility.

The Engage Model is a chronic care approach to support hearing loss self-management of ARHL. Engage includes (a) hearing screening for all residents, (b) an individualized communication plan for those with an identified hearing loss (e.g., one-to-one, group, telephone, television plans, hearing aid trouble shooting, communication strategies, etc.), (c) provision of simple, non-custom amplifiers, (d) referral to audiology if needed, and (e) ongoing support provided by trained personnel (Communication Facilitator) under the supervision of the audiologist.

DETAILED DESCRIPTION:
The study is employing an open cohort stepped-wedge cluster randomized design with a phased, randomized roll out. The stepped wedge design is a useful design for the evaluation of complex health care interventions particularly when the intervention is believed to be beneficial with minimal risk. This design is increasingly being used to evaluate interventions involving health care delivery and has several advantages:

1. allowing the clinical teams to roll out the intervention in a small number of facilities in a timely, systematic manner (interventions are not part of the research protocol)
2. possibly increasing participation and buy-in since all facilities will eventually implement the intervention during the study
3. possible increase in statistical power compared to a cluster randomized trial due to increase in data collection and within cluster comparisons.

Our intervention is applied at the facility level (cluster) but the primary outcomes are obtained at the resident level. In this open cohort design, all residents in a facility are identified to participate but some may leave the facility and others will move into the facility over the course of the study. The interventions are standard care at UPMC and are at the facility and individual level regardless of participation in the research project by any individual.

The 10 facilities participating in the study all currently receive the Consult Model of care. These same facilities are targeted to receive the Engage Model of care over the next three years as part of the standard care in these facilities. Residents enrolled in the study during any time period will be followed until the end of the study or until they are no longer a resident of the facility, whichever comes first. This implies that crossover to the intervention is not only at the facility level but also the resident level. Once the intervention is available at a facility, residents will be exposed to the intervention continuously regardless of enrollment for the study measures. The resident level outcomes of satisfaction with social participation and hearing-specific HRQoL will be measured every 5 months for the duration of the study. In addition, staff satisfaction and family burden will be surveyed every 5 months.

NOTE: The clinicaltrials.gov record was updated after data collection ended to correct the study arms and interventions. The study arms were originally and incorrectly documented in clinicaltrials.gov as the resident, caregiver, and staff cohorts rather than the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate and
* Being a resident, staff member or family member of a resident at one of the participating Assisted Living/Personal Care Facilities.

Exclusion Criteria:

* Unwillingness to participate
* Not being a Resident, staff member or family member of a resident at one of eight Assisted Living/Personal Care Facilities.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Palmer, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data, including protocol, statistical analysis and full data set may be shared with investigators conducting similar research or for educational purposes. No identifiable data will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available after the conclusion of the study and will be available
Access Criteria: Access to the data will be determined by the PIs and funding agency (PCORI). Requests for the data can be made to them and will be considered before dissemination.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was an open cohort stepped wedge design with continuous recruitment and enrollment. Residents were enrolled at Time Period 0 but could be enrolled at any time period of the study due to being a new resident of the facility or being interested at the time period they were approached. The protocol enrollment reflects the total number enrolled at all 10 facilities across 6 time points (Time Periods 0-5).
Pre-assignment Details: Available family members of residents in the study and staff in the facilities were asked to complete surveys for the secondary outcomes during each data collection period. These individuals were not tracked across time periods or documented for lost-to-follow-up or discontinuation from the study. The number of surveys and the corresponding results are presented in the secondary outcomes. No adverse event data were required to be collected for family members and staff.
Units Other Than Participants: residential facility
Groups:
- Group 1 (HearCARE Start at T1): Facilities had the Consult Model for Time Period 0 then started the HearCARE program at Time Period 1 and continued with the HearCARE program through Time Period 5.
- Group 2 (HearCARE Start at T2): Facilities had the Consult Model for Time Periods 0 and 1 then started the HearCARE program at Time Period 2 and continued with the HearCARE program through Time Period 5.
- Group 3 (HearCARE Start at T3): Facilities had the Consult Model for Time Periods 0, 1 and 2 then started the HearCARE program at Time Period 3 and continued with the HearCARE program through Time Period 5.
- Group 4 (HearCARE Start at T4): Facilities had the Consult Model for Time Periods 0, 1, 2, and 3 then started the HearCARE program at Time Period 4 and continued with the HearCARE program through Time Period 5.
- Group 5 (HearCARE Start at T5): Facilities had the Consult Model for Time Periods 0-4 then started the HearCARE program at Time Period 5.
Period: Time Period 0
Arm/Group | Group 1 (HearCARE Start at T1) | Group 2 (HearCARE Start at T2) | Group 3 (HearCARE Start at T3) | Group 4 (HearCARE Start at T4) | Group 5 (HearCARE Start at T5)
Started | 62; 2 residential facility | 55; 2 residential facility | 87; 2 residential facility | 77; 2 residential facility | 44; 2 residential facility
Completed | 47; 2 residential facility | 49; 2 residential facility | 68; 2 residential facility | 68; 2 residential facility | 36; 2 residential facility
Not Completed | 15; 0 residential facility | 6; 0 residential facility | 19; 0 residential facility | 9; 0 residential facility | 8; 0 residential facility
Not completed — Discontinued due to death or moving to higher level of care | 15 | 6 | 19 | 9 | 8
Period: Time Period 1
Arm/Group | Group 1 (HearCARE Start at T1) | Group 2 (HearCARE Start at T2) | Group 3 (HearCARE Start at T3) | Group 4 (HearCARE Start at T4) | Group 5 (HearCARE Start at T5)
Started | 69; 2 residential facility | 84; 2 residential facility | 89; 2 residential facility | 87; 2 residential facility | 58; 2 residential facility
Completed | 55; 2 residential facility | 67; 2 residential facility | 79; 2 residential facility | 69; 2 residential facility | 42; 2 residential facility
Not Completed | 14; 0 residential facility | 17; 0 residential facility | 10; 0 residential facility | 18; 0 residential facility | 16; 0 residential facility
Not completed — Missing follow up | 1 | 3 | 1 | 3 | 2
Not completed — Discontinued due to death or moving to higher level of care | 13 | 14 | 9 | 15 | 14
Period: Time Period 2
Arm/Group | Group 1 (HearCARE Start at T1) | Group 2 (HearCARE Start at T2) | Group 3 (HearCARE Start at T3) | Group 4 (HearCARE Start at T4) | Group 5 (HearCARE Start at T5)
Started | 75; 2 residential facility | 75; 2 residential facility | 99; 2 residential facility | 80; 2 residential facility | 51; 2 residential facility
Completed | 59; 2 residential facility | 59; 2 residential facility | 72; 2 residential facility | 65; 2 residential facility | 42; 2 residential facility
Not Completed | 16; 0 residential facility | 16; 0 residential facility | 27; 0 residential facility | 15; 0 residential facility | 9; 0 residential facility
Not completed — Missing follow up | 1 | 8 | 7 | 0 | 1
Not completed — Discontinued due to death or moved to higher level of care | 15 | 8 | 20 | 15 | 8
Period: Time Period 3
Arm/Group | Group 1 (HearCARE Start at T1) | Group 2 (HearCARE Start at T2) | Group 3 (HearCARE Start at T3) | Group 4 (HearCARE Start at T4) | Group 5 (HearCARE Start at T5)
Started | 87; 2 residential facility | 82; 2 residential facility | 96; 2 residential facility | 65; 2 residential facility | 56; 2 residential facility
Completed | 74; 2 residential facility | 72; 2 residential facility | 81; 2 residential facility | 59; 2 residential facility | 53; 2 residential facility
Not Completed | 13; 0 residential facility | 10; 0 residential facility | 15; 0 residential facility | 6; 0 residential facility | 3; 0 residential facility
Not completed — Missing follow up | 8 | 6 | 4 | 3 | 0
Not completed — Discontinued due to death or moved to higher level of care | 5 | 4 | 11 | 3 | 3
Period: Time Period 4
Arm/Group | Group 1 (HearCARE Start at T1) | Group 2 (HearCARE Start at T2) | Group 3 (HearCARE Start at T3) | Group 4 (HearCARE Start at T4) | Group 5 (HearCARE Start at T5)
Started | 96; 2 residential facility | 92; 2 residential facility | 100; 2 residential facility | 70; 2 residential facility | 62; 2 residential facility
Completed | 77; 2 residential facility | 86; 2 residential facility | 87; 2 residential facility | 67; 2 residential facility | 52; 2 residential facility
Not Completed | 19; 0 residential facility | 6; 0 residential facility | 13; 0 residential facility | 3; 0 residential facility | 10; 0 residential facility
Not completed — Missing follow up | 17 | 3 | 4 | 2 | 1
Not completed — Discontinued due to death or moved to higher level of care | 2 | 3 | 9 | 1 | 9
Period: Time Period 5
Arm/Group | Group 1 (HearCARE Start at T1) | Group 2 (HearCARE Start at T2) | Group 3 (HearCARE Start at T3) | Group 4 (HearCARE Start at T4) | Group 5 (HearCARE Start at T5)
Started | 112; 2 residential facility | 98; 2 residential facility | 97; 2 residential facility | 80; 2 residential facility | 59; 2 residential facility
Completed | 101; 2 residential facility | 90; 2 residential facility | 85; 2 residential facility | 77; 2 residential facility | 48; 2 residential facility
Not Completed | 11; 0 residential facility | 8; 0 residential facility | 12; 0 residential facility | 3; 0 residential facility | 11; 0 residential facility
Not completed — Missing follow up | 11 | 8 | 12 | 3 | 11

BASELINE CHARACTERISTICS:
Population: Residents who were ever enrolled into the study over the all time periods (Time Period 0 through Time Period 5) of the stepped wedge cluster randomized trial.
Groups:
- Group 1 (HearCARE Start T1): Participants in these facilities had the Consult Model for Time Period 0 then started the HearCARE program at Time Period 1 and continued with the HearCARE program through Time Period 5.
- Group 2 (HearCARE Start T2): Participants in these facilities had the Consult Model for Time Periods 0 and 1 then started the HearCARE program at Time Period 2 and continued with the HearCARE program through Time Period 5.
- Group 3 (HearCARE Start T3): Participants in these facilities had the Consult Model for Time Periods 0, 1 and 2 then started the HearCARE program at Time Period 3 and continued with the HearCARE program through Time Period 5.
- Group 4 (HearCARE Start T4): Participants in these facilities had the Consult Model for Time Periods 0, 1, 2, and 3 then started the HearCARE program at Time Period 4 and continued with the HearCARE program through Time Period 5.
- Group 5 (HearCARE Start T5): Participants in these facilities had the Consult Model for Time Periods 0-4 then started the HearCARE program at Time Period 5.
- Total: Total of all reporting groups
Arm/Group | Group 1 (HearCARE Start T1) | Group 2 (HearCARE Start T2) | Group 3 (HearCARE Start T3) | Group 4 (HearCARE Start T4) | Group 5 (HearCARE Start T5) | Total
Number analyzed (Participants) | 162 | 133 | 165 | 123 | 101 | 684
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Analysis for those with information on age. Some participants did not complete this information.
  years
    number analyzed (Participants) | 147 | 106 | 151 | 110 | 86 | 600
    (all) | 89.3 (7.8) | 87.8 (7.1) | 87.3 (8.3) | 89.0 (8.4) | 83.8 (8.6) | 87.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 96 | 126 | 89 | 61 | 495
  Male | 39 | 37 | 39 | 34 | 40 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 161 | 133 | 165 | 123 | 101 | 683
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Self-reported race
  participants
    White | 155 | 120 | 160 | 116 | 92 | 643
    Not White | 4 | 6 | 3 | 2 | 0 | 15
    Not Reported | 3 | 7 | 2 | 5 | 9 | 26
Region of Enrollment [Number; unit: participants]
  United States | 162 | 133 | 165 | 123 | 101 | 684
Hearing Handicap Inventory at Enrollment [Mean (Standard Deviation); unit: units on a scale] — Hearing Handicap Inventory for the Elderly captures social and emotional hearing handicap. 10 items with responses scored 0, 2, and 4 for 'No', 'Sometimes', and 'Yes'; min total score is 0 and maximum is 40. Higher scores indicate worse impact of hearing difficulties on activities and participation. Population: Analysis among those with survey information. Some participants did not complete the survey.
  units on a scale
    number analyzed (Participants) | 159 | 131 | 162 | 115 | 98 | 665
    (all) | 8.2 (9.2) | 9.0 (9.0) | 8.6 (8.9) | 8.0 (9.5) | 6.5 (8.4) | 8.2 (9.0)
PROMIS Participation at Enrollment [Mean (Standard Deviation); unit: T-score] — PROMIS Satisfaction with Participation in Discretionary Social Activities SF7a self-reported contentment with leisure interests and relationships with friends. T- scores are provided ranging from 27 to 65.6 where higher scores indicate more satisfaction (50 indicates the population mean with a standard deviation of 10). Population: Analysis of those with survey data. Some participants did not complete the survey.
  T-score
    number analyzed (Participants) | 151 | 117 | 159 | 113 | 98 | 638
    (all) | 49.4 (7.1) | 50.6 (8.1) | 49.9 (8.8) | 48.1 (7.2) | 49.8 (7.3) | 49.6 (7.8)
Pure tone average right side [Mean (Standard Deviation); unit: decibels] — Indication of hearing ability in the right ear. Average of the threshold at 500, 1000, and 2000 Hz. Threshold is the lowest (quietest) level at which an individual can detect a sound. The average is a good estimate of severity of loss related to hearing speech (those frequencies are important to speech). The minimum is 0 dB HL (best) and the maximum is 90 dB HL (worst). Small numbers represent better hearing, higher number represents more hearing loss. Population: Analysis conducted for participants with hearing assessments.
  decibels
    number analyzed (Participants) | 121 | 69 | 117 | 64 | 83 | 454
    (all) | 43.5 (14.2) | 47.0 (15.8) | 44.1 (17.5) | 47.6 (17.0) | 39.5 (14.0) | 44.0 (15.9)
Pure tone average left side [Mean (Standard Deviation); unit: decibels] — Indication of hearing ability in the left ear. Average of the threshold at 500, 1000, and 2000 Hz. Threshold is the lowest (quietest) level at which an individual can detect a sound. The average is a good estimate of severity of loss related to hearing speech (those frequencies are important to speech). The minimum is 0 dB HL (best) and the maximum is 90 dB HL (worst). Small numbers represent better hearing, higher number represents more hearing loss. Population: Analysis among those with hearing assessments.
  decibels
    number analyzed (Participants) | 122 | 70 | 115 | 63 | 83 | 453
    (all) | 43.6 (14.8) | 47.3 (15.8) | 44.1 (17.0) | 47.0 (14.9) | 40.7 (14.3) | 44.3 (15.6)

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction With Social Participation
Description: PROMIS Satisfaction with Participation in Discretionary Social Activities SF7a self-reported contentment with leisure interests and relationships with friends. T- scores are provided ranging from 27 to 65.6 where higher scores indicate more satisfaction (50 indicates the population mean with a standard deviation of 10).
Time Frame: Baseline (T0), at 5 (T1), 10 (T2), 15 (T3), 20 (T4) and 25 (T5) months
Population: The overall number of participants analyzed represents the number of unique participants who provided data across the time points. The number at each time point represents the number of participants who contributed survey data at that time point. Due to the open cohort nature of the trial, the number with survey data represents both those enrolled who did not leave the cohort and those with survey data entering the cohort (newly enrolled).
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Group 1 (HearCARE Start at T1) | Group 2 (HearCARE Start at T2) | Group 3 (HearCARE Start at T3) | Group 4 (HearCARE Start at T4) | Group 5 (HearCARE Start at T5)
Number analyzed (Participants) | 162 | 133 | 165 | 123 | 101
T-score
  Baseline (Time 0): number analyzed (Participants) | 53 | 53 | 85 | 69 | 43
  Baseline (Time 0) | 49.7 (7.9) | 52.8 (8.9) | 51.2 (10.3) | 49.4 (6.6) | 51.7 (7.6)
  5 months (Time 1): number analyzed (Participants) | 60 | 59 | 84 | 79 | 54
  5 months (Time 1) | 49.7 (7.8) | 48.4 (6.7) | 47.6 (8.7) | 48.1 (5.6) | 48.1 (7.0)
  10 months (Time 2): number analyzed (Participants) | 72 | 55 | 81 | 76 | 45
  10 months (Time 2) | 48.1 (7.1) | 47.6 (6.1) | 49.4 (7.0) | 48.6 (7.0) | 47.4 (6.0)
  15 months (Time 3): number analyzed (Participants) | 73 | 60 | 68 | 50 | 52
  15 months (Time 3) | 52.0 (7.1) | 47.1 (6.5) | 45.4 (6.2) | 49.9 (8.1) | 48.4 (6.6)
  20 months (Time 4): number analyzed (Participants) | 54 | 66 | 72 | 53 | 57
  20 months (Time 4) | 49.4 (5.6) | 49.0 (7.1) | 47.2 (6.3) | 48.1 (6.8) | 48.2 (6.4)
  25 months (Time 5): number analyzed (Participants) | 59 | 67 | 56 | 61 | 41
  25 months (Time 5) | 49.1 (7.3) | 48.2 (7.8) | 49.6 (8.2) | 47.4 (7.2) | 48.9 (6.7)
Statistical Analysis 1: Comparison: Group 1 (HearCARE Start at T1) vs Group 2 (HearCARE Start at T2) vs Group 3 (HearCARE Start at T3) vs Group 4 (HearCARE Start at T4) vs Group 5 (HearCARE Start at T5); The null hypothesis is that the HearCARE intervention does not improve satisfaction with social participation; Test type: Superiority; p = 0.58, Mixed Models Analysis; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-1.10 to 1.96] — Difference in the adjusted means for the Consult model and HearCARE model

2. Primary Outcome: Hearing-Specific Health-Related Quality of Life
Description: Hearing Handicap Inventory for the Elderly captures social and emotional hearing handicap. 10 items with responses scored 0, 2, and 4 for 'No', 'Sometimes', and 'Yes'; min total score is 0 and maximum is 40. Higher scores indicate worse impact of hearing difficulties on activities and participation.
Time Frame: Baseline, at 5, 10, 15, 20 and 25 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (HearCARE Start at T1) | Group 2 (HearCARE Start at T2) | Group 3 (HearCARE Start at T3) | Group 4 (HearCARE Start at T4) | Group 5 (HearCARE Start at T5)
Number analyzed (Participants) | 162 | 133 | 165 | 123 | 101
score on a scale
  Baseline (Time 0): number analyzed (Participants) | 60 | 55 | 86 | 71 | 43
  Baseline (Time 0) | 10.2 (11.2) | 10.6 (9.6) | 9.2 (10.2) | 7.5 (8.9) | 8.1 (9.4)
  5 months (Time 1): number analyzed (Participants) | 66 | 75 | 83 | 79 | 55
  5 months (Time 1) | 9.4 (9.6) | 10.9 (10.1) | 9.4 (9.2) | 9.2 (10.9) | 8.9 (9.1)
  10 months (Time 2): number analyzed (Participants) | 73 | 54 | 83 | 76 | 45
  10 months (Time 2) | 8.9 (8.8) | 11.6 (10.2) | 8.9 (8.5) | 9.2 (9.0) | 5.6 (7.0)
  15 months (Time 3): number analyzed (Participants) | 74 | 61 | 69 | 54 | 52
  15 months (Time 3) | 7.3 (8.9) | 9.8 (10.0) | 9.5 (9.2) | 10.1 (9.5) | 6.7 (8.5)
  20 months (Time 4): number analyzed (Participants) | 54 | 68 | 73 | 54 | 57
  20 months (Time 4) | 6.9 (8.3) | 8.5 (8.3) | 7.9 (7.7) | 9.7 (8.9) | 7.0 (8.8)
  25 months (Time 5): number analyzed (Participants) | 69 | 66 | 58 | 57 | 43
  25 months (Time 5) | 9.0 (11.0) | 8.5 (10.0) | 4.4 (5.0) | 6.9 (8.5) | 5.6 (8.6)
Statistical Analysis 1: Comparison: Group 1 (HearCARE Start at T1) vs Group 2 (HearCARE Start at T2) vs Group 3 (HearCARE Start at T3) vs Group 4 (HearCARE Start at T4) vs Group 5 (HearCARE Start at T5); The null hypothesis is that the HearCARE intervention does not improve hearing related quality of life; Test type: Superiority; p = 0.95, Mixed Models Analysis; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-1.13 to 1.10] — The estimated parameter represents the difference between the adjusted means for the Consult and HearCARE models

3. Secondary Outcome: Family Burden
Description: Zarit Burden Interview is a 4-item questionnaire that measures caregiver burden. The 4 items each have responses ranging from 0='Never' to 4='Nearly Always'. Item responses are summed to produce the total score that ranges from 0 to 16 with higher scores indicating more burden.
Time Frame: Baseline, at 5, 10, 15, 20 and 25 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (HearCARE Start at T1) | Group 2 (HearCARE Start at T2) | Group 3 (HearCARE Start at T3) | Group 4 (HearCARE Start at T4) | Group 5 (HearCARE Start at T5)
Number analyzed (Participants) | 78 | 85 | 116 | 83 | 72
score on a scale
  Baseline (Time 0): number analyzed (Participants) | 30 | 29 | 55 | 32 | 30
  Baseline (Time 0) | 5.5 (3.7) | 4.4 (3.4) | 5.4 (3.0) | 4.7 (3.6) | 4.9 (3.0)
  5 months (Time 1): number analyzed (Participants) | 21 | 37 | 38 | 30 | 26
  5 months (Time 1) | 3.6 (2.8) | 3.9 (2.9) | 4.5 (3.1) | 4.2 (3.7) | 4.6 (3.4)
  10 months (Time 2): number analyzed (Participants) | 17 | 31 | 56 | 28 | 14
  10 months (Time 2) | 3.9 (2.8) | 6.7 (4.4) | 5.6 (3.3) | 4.8 (3.7) | 4.8 (3.8)
  15 months (Time 3): number analyzed (Participants) | 15 | 12 | 40 | 27 | 22
  15 months (Time 3) | 5.1 (3.7) | 5.2 (4.6) | 5.4 (3.0) | 4.1 (3.8) | 5.0 (4.8)
  20 months (Time 4): number analyzed (Participants) | 8 | 5 | 38 | 23 | 22
  20 months (Time 4) | 4.8 (2.8) | 3 (2.8) | 5.9 (3.7) | 5.0 (3.5) | 5.3 (3.9)
  25 months (Time 5): number analyzed (Participants) | 21 | 20 | 26 | 10 | 16
  25 months (Time 5) | 5.1 (2.7) | 4.3 (4.0) | 5.4 (2.8) | 4.6 (3.9) | 4.4 (3.6)
Statistical Analysis 1: Comparison: Group 1 (HearCARE Start at T1) vs Group 2 (HearCARE Start at T2) vs Group 3 (HearCARE Start at T3) vs Group 4 (HearCARE Start at T4) vs Group 5 (HearCARE Start at T5); Test type: Superiority; p = 0.96, Mixed Models Analysis; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-1.20 to 1.14] — Estimated Value represents the difference in the means for the Consult and HearCARE models

4. Secondary Outcome: Staff Satisfaction
Description: Michigan Organizational Assessment Questionnaire (MOAQ) is a 3-item questionnaire that measures satisfaction with one's job. Items have responses ranging from 1='Agree Strongly' to 6='Disagree Strongly'. The combined score is the average of the 3 items with one item reverse scored. Higher scores indicate less satisfaction.
Time Frame: Baseline, at 5, 10, 15, 20 and 25 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 (HearCARE Start at T1) | Group 2 (HearCARE Start at T2) | Group 3 (HearCARE Start at T3) | Group 4 (HearCARE Start at T4) | Group 5 (HearCARE Start at T5)
Number analyzed (Participants) | 130 | 83 | 138 | 70 | 81
score on a scale
  Baseline (Time 0): number analyzed (Participants) | 17 | 4 | 35 | 19 | 20
  Baseline (Time 0) | 2.1 (1.0) | 1.3 (0.5) | 1.6 (0.8) | 2.1 (1.0) | 1.8 (0.6)
  5 months (Time 1): number analyzed (Participants) | 42 | 55 | 46 | 17 | 20
  5 months (Time 1) | 1.9 (1.0) | 1.9 (0.8) | 1.6 (0.7) | 1.8 (0.9) | 1.8 (0.7)
  10 months (Time 2): number analyzed (Participants) | 31 | 9 | 55 | 10 | 2
  10 months (Time 2) | 1.7 (0.8) | 1.1 (0.3) | 2.2 (1.2) | 1.4 (0.5) | 1.7 (0)
  15 months (Time 3): number analyzed (Participants) | 40 | 8 | 40 | 16 | 18
  15 months (Time 3) | 1.8 (0.8) | 1.3 (0.6) | 2.0 (1.0) | 1.7 (0.8) | 2.1 (0.9)
  20 months (Time 4): number analyzed (Participants) | 37 | 12 | 35 | 18 | 27
  20 months (Time 4) | 1.8 (1.1) | 1.5 (0.8) | 1.9 (1.1) | 1.4 (0.6) | 1.8 (0.8)
  25 months (Time 5): number analyzed (Participants) | 38 | 12 | 36 | 15 | 26
  25 months (Time 5) | 1.6 (0.8) | 1.4 (0.7) | 1.7 (0.7) | 1.4 (0.5) | 1.9 (0.8)
Statistical Analysis 1: Comparison: Group 1 (HearCARE Start at T1) vs Group 2 (HearCARE Start at T2) vs Group 3 (HearCARE Start at T3) vs Group 4 (HearCARE Start at T4) vs Group 5 (HearCARE Start at T5); Test type: Superiority; p = 0.13, Mixed Models Analysis; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.07 to 0.48] — The Estimated Value is the difference between the means of the Consult and HearCARE models

ADVERSE EVENTS:
Time Frame: 25 months from study start (Time Point 0 through Time Point 5)
Description: This study was considered exempt from collecting data on adverse events due to the nature of the intervention and the data being collected. Deaths were recorded but not required to be documented as serious adverse events per the Institutional Review Board.
Groups:
- Group 1 (2 Residential Facilities): Participants in these facilities had the Consult Model for Time Period 0 then started the HearCARE program at Time Period 1 and continued with the HearCARE program through Time Period 5.
- Group 2 (2 Residential Facilities): Participants in these facilities had the Consult Model for Time Periods 0 and 1 then started the HearCARE program at Time Period 2 and continued with the HearCARE program through Time Period 5.
- Group 3 (2 Residential Facilities): Participants in these facilities had the Consult Model for Time Periods 0, 1 and 2 then started the HearCARE program at Time Period 3 and continued with the HearCARE program through Time Period 5.
- Group 4 (2 Residential Facilities): Participants in these facilities had the Consult Model for Time Periods 0, 1, 2, and 3 then started the HearCARE program at Time Period 4 and continued with the HearCARE program through Time Period 5.
- Group 5 (2 Residential Facilities): Participants in these facilities had the Consult Model for Time Periods 0-4 then started the HearCARE program at Time Period 5.
Arm/Group | Group 1 (2 Residential Facilities) | Group 2 (2 Residential Facilities) | Group 3 (2 Residential Facilities) | Group 4 (2 Residential Facilities) | Group 5 (2 Residential Facilities)
All-Cause Mortality (participants affected / at risk) | 25/162 | 23/133 | 53/165 | 20/123 | 24/101
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT04575051/Prot_SAP_000.pdf